CLINICAL TRIAL: NCT01736956
Title: Fetal Intervention for Aortic Stenosis and Evolving Hypoplastic Left Heart Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-08688
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Aortic Stenosis; Hypoplastic Left Heart Syndrome
Keywords: aortic stenosis; hypoplastic left heart syndrome; fetal aortic valvuloplasty
MeSH Terms: conditions — Aortic Valve Stenosis; Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fetal Aortic Valvuloplasty (Experimental): Subjects will undergo fetal aortic valvuloplasty
  Interventions: Procedure: Fetal Aortic Valvuloplasty
- Control (No Intervention): Control group. Will receive standard prenatal and postnatal care.

INTERVENTIONS:
Procedure: Fetal Aortic Valvuloplasty — Fetuses in the intervention group will undergo in utero balloon aortic valvuloplasty via a transuterine, perventricular approach. Fetuses in the control group will have no invasive intervention while in utero.
  Other Names: Fetal balloon aortic valvuloplasty
  Arms: Fetal Aortic Valvuloplasty

SUMMARY:
For fetuses with severe aortic stenosis, in utero balloon aortic valvuloplasty may improve fetal growth of left heart structures and thus improve potential for biventricular repair strategies after birth.

DETAILED DESCRIPTION:
Fetal aortic stenosis is an anatomically simple birth defect in which there is partial blockage of the aortic valve, limiting blood flow out of the left side of the heart. If the blockage becomes severe in fetal life, the left heart structures may stop growing and the baby may be born with hypoplastic left heart syndrome (HLHS), a lethal condition without neonatal heart surgery or heart transplantation. Standard treatment for babies born with HLHS includes three major cardiac operations before the age of 6 years. Postnatal outcomes for HLHS are uncertain and vary with patient; however, the few adult survivors are currently suffering substantial medical problems, including a high incidence of neurologic problems. For fetuses with severe obstruction, fetal intervention may improve outcomes by increasing flow through the left heart, thus improving left heart function and encouraging continued growth of the left heart structures. If fetal intervention can preserve left heart function and growth, this should provide a better prognosis for the baby and allow for biventricular repair strategies after birth.

This research study is a prospective, non-randomized clinical trial of 30 patients that will assess the safety and efficacy of in utero percutaneous balloon dilation of fetal aortic valve with severe stenosis. This technique has been successfully used to perform postnatal aortic valve dilations for several decades, but has had limited application and study in utero.

Pregnant women carrying a fetus diagnosed with severe aortic stenosis will be referred to the University of California, San Francisco Fetal Treatment Center for evaluation, initial screening and counseling. If all fetal and maternal inclusion criteria are met, the balloon aortic valvuloplasty operation will be offered to the pregnant woman. Patients who do not meet study eligibility or decline prenatal intervention will be offered the option to enroll as a study control.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman carrying a fetus with normal cardiac segmental anatomy and severe aortic stenosis as defined by:

  * Dysplastic/stenotic aortic valve with forward flow, with or without gradient, and no significant insufficiency
  * If mitral insufficiency (incomplete closure of the mitral valve)is present, left ventricle systolic pressure calculation must be ≥ a normal systemic blood pressure (BP) for gestational age
  * Retrograde aortic arch flow
  * Left to right atrial shunting
  * Left ventricle length no less than 90% the length of the right ventricle
* Maternal age ≥ 16 years of age;
* Gestational age: 17 0/7-30 6/7 weeks' gestation as determined by clinical information and evaluation of first ultrasound. (Aortic valve dilation procedure cannot be performed until 18 0/7 weeks);
* Normal karyotype with written confirmation of results. Results by fluorescence in situ hybridization (FISH) for aneuploidy will be acceptable if the patient is at 24 weeks or more; non-invasive testing is acceptable (maternal serum testing for cell-free fetal DNA, currently commercially available).
* Singleton pregnancy;
* Able to travel to study site for study evaluation, procedures, and visits;
* Support person to travel and stay with patient (support person will be required to sign the support person consent form);
* Has received pre-authorization for insurance for fetal intervention or has the ability to self-pay for study treatment

Exclusion Criteria:

* Failure to meet all inclusion criteria;
* Multi-fetal pregnancy;
* Insulin dependent pregestational diabetes;
* Fetal anomaly not related to aortic stenosis. A detailed fetal anatomic ultrasound will be conducted before consideration for the study and if the finding is abnormal, the patient will be excluded;
* Current or planned cerclage or documented history of incompetent cervix;
* Placenta previa or placental abruption;
* Short cervix (< 20mm) measured by cervical ultrasound;
* Previous spontaneous delivery prior to 37 weeks of a singleton pregnancy. If the study candidate had intact membranes and was induced, this is not considered spontaneous. Stillbirths prior to 37 weeks are not exclusionary.
* Obesity as defined by body mass index of 35 or greater;
* Maternal-fetal Rh isoimmunization, Kell sensitization or a history of neonatal alloimmune thrombocytopenia;
* Positive maternal HIV status. This is due to the increased risk of transmission to the fetus during the maternal-fetal procedure. If the patient's HIV status is unknown, the patient must be tested and found to have negative results before she can be entered into the fetal treatment group;
* Known Hepatitis C positivity. If the patient's Hepatitis C status is unknown, she does not need to be screened;
* Other maternal medical condition which is a contraindication to surgery or general anesthesia, such as asthma, cardiac disease, the refusal of a blood transfusion, or a previous hysterotomy in the active segment of the uterus;
* Patient does not have a support person (e.g., husband, partner, mother), or that support person is unwilling to sign the support person consent form;
* Inability to comply with the travel and follow-up requirements of the study;
* Patient does not meet other psychosocial criteria to handle the implications of the study;
* Participation in another intervention study that influences maternal and fetal morbidity and mortality;
* Maternal hypertension which would increase the risk of preeclampsia or preterm delivery (including, but not limited to: uncontrolled hypertension, chronic hypertension with end organ damage and new onset hypertension in current pregnancy).

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-10; Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Improved fetal mitral valve and left ventricular growth | Monthly until birth, and after birth until three years of age
  The primary outcome variable is fetal mitral valve and left ventricular growth due to successful balloon dilation, as determined by serial echocardiographic measurements

SECONDARY OUTCOMES:
Neonatal survival at 365 days of life | 365 days after birth

OTHER OUTCOMES:
Neurodevelopmental and functional status | Birth to 30 months
  Neurodevelopmental and functional status at 12 and 30 months of life, as determined by physical exam, echocardiogram, neuro-developmental testing, and hearing testing.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Moon-Grady, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco Fetal Treatment Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No